CLINICAL TRIAL: NCT06740669
Title: Effects of VE, Focus, Expressive Touch on Pain, Anxiety, Breastfeeding and Mobilization in Women Delivering by Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mine Gokduman Keles, Asst.Prof. Mine GÖKDUMAN KELEŞ PhD.MİDW,FERY, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 05.11.2024 _ 2024/11 GO 202
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Women; Postnatal Care
Keywords: Virtual reality,; Focus; Expressive touch; Pain; Anxiety; Breastfeeding
MeSH Terms: conditions — Pain; Anxiety Disorders; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Women in the control group will receive routine care and breastfeeding support will be provided to these women.
- Virtual reality glasses (VR) application (Active Comparator)
  Interventions: Behavioral: Virtual reality glasses (VR) application
- Expressive touch applications (Active Comparator)
  Interventions: Behavioral: Those who are applied expressive touch
- Focusing (Active Comparator)
  Interventions: Behavioral: Focus

INTERVENTIONS:
Behavioral: Virtual reality glasses (VR) application — It will be evaluated at 1 and 6 hours after the Caesarean section and a relaxing video called Relaxation (https://www.youtube.com/watch?v=H1iboKia3AQ, a video containing nature scenes accompanied by nature sounds) will be shown for a maximum of 20 minutes through virtual reality glasses (Toker and Gökduman Keleş, 2024).
  Arms: Virtual reality glasses (VR) application
Behavioral: Those who are applied expressive touch — Expressive touch does not require any preparation other than warming the hands to the same temperature as the body temperature. During expressive touch practice; the parts of the body that are touched the most are the hands, arms, forehead, hair and shoulders. The hands are massaged during the touch and the arms and shoulders are lightly touched before and after the massage, so that the expressive touch made on the hands is effective (Pinar and Demirel, 2021; Routasalo, 1999) After the evaluation, the researcher will apply expressive touch to one of the mother's hands for an average of 15-20 minutes
  Arms: Expressive touch applications
Behavioral: Focus — . The researcher mother will be asked to focus on her baby for 10 minutes (Kiliçli Id and Zeyneloglu Id, 2024; Vamour et al., 2019).
  Arms: Focusing

SUMMARY:
Cesarean section is one of the most common surgical interventions in many countries. It is seen that 21.1% of women worldwide, 57.5% in Turkey, give birth by cesarean section. 99.6% of women have pain in the first 24 hours after cesarean section and oral analgesia is not sufficient for pain. It is seen that pain has an effect on recovery and breastfeeding after CS.This study will be conducted to determine the effects of non-pharmacological methods, virtual reality glasses, focusing and expressive touch on pain, anxiety, breastfeeding and mobilization in women giving birth by cesarean section. The ınvestigators aim to contribute to the midwifery and nursing care literature with the findings and results of the study.

DETAILED DESCRIPTION:
Subject: Cesarean section is one of the most common surgical interventions in many countries. It is observed that 21.1% of women worldwide and 57.5% in Turkey give birth by cesarean section. 99.6% of women have pain in the first 24 hours after cesarean section and oral analgesia is not sufficient for pain . Pain is observed to have an effect on recovery and breastfeeding after CS . In the literature, it has been reported that some applications such as acupressure, acupuncture, relaxation exercises, foot reflexology, aromatherapy, music, transcutaneous electrical nerve stimulation, and distraction, which are non-pharmacological methods in the adjunctive treatment of postoperative pain, reduce pain, fatigue, and anxiety, accelerate mobilization, and positively affect breastfeeding .. In general, non-pharmacological methods significantly affect pain after cesarean section . Based on these studies, it is seen that non-pharmacological methods applied to reduce anxiety and pain after cesarean section are effective. In recent years, virtual reality glasses (VR) , focusing and expressive touching have taken their place in the literature. When the literature is examined, it is seen that virtual reality glasses, focus and expressive touch reduce the pain level and provide anxiety reduction.

No study has been found on the application of virtual reality glasses, focus and expressive touch in reducing pain and anxiety after cesarean section. This study will be conducted to determine the effects of virtual reality glasses, focus and expressive touch, which are non-pharmacological methods, on pain, anxiety, breastfeeding and mobilization in women who give birth by cesarean section.

The ınvestigators aim for the findings and results of the study to contribute to the midwifery and nursing care literature.

ELIGIBILITY:
Inclusion Criteria:

- Women who do not have any psychiatric illness,

* Those who do not have any vision, hearing or perception problems,
* Those who do not have any communication problems (can speak Turkish),
* Those who accept to participate in the study verbally and in writing were included in the study.
* Those who are between the ages of 18-35,
* Those who have had a singleton birth,
* Those who have had the operation with regional anesthesia (spinal or epidural anesthesia),

Exclusion Criteria:

* Exclusion Criteria from the Study

  * Receiving controlled analgesia after cesarean section
  * Having a psychiatric diagnosis such as anxiety and depression
  * Those who develop postpartum complications
  * Women who want to leave the study at any stage of the study will be excluded from the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 208 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 1 HOUR
  The numerical pain rating scale (NAS) is used to assess anxiety severity. In the numerical rating scale, anxiety is between 0 and 10 points.
VAS Anxiety | 1 HOUR
  The numerical pain rating scale (PAS) is used to assess anxiety severity. Anxiety is rated between 0 and 10 points on the numerical rating scale
Mobilization | 6HOUR
  The decision to start or continue mobilization will be made by the healthcare professional working in the clinic.
  The mobilization status of the women will be evaluated. The examiner will note the success or failure of the patient's mobilization along with its duration. (the beginning of the measurement was determined as the moment the patient got up from the sitting position and the end of the measurement was determined as the moment the patient returned to the bed). If the patient got up from the bed and started walking (took at least one step), they received a score of 1 (successful) on the questionnaire form. If they got up but did not take a single step while returning to the sitting position, they received a score of 0. The mobilization time will be measured in minutes
6-Minute Walking Test (6MWT) | 6 HOUR
  6MWT will be used to evaluate the physical functions of patients. During this test, a 30-meter track with a hard surface will be walked at a normal pace for six minutes. This track is marked every 3 meters and a cone is placed at the end of this 30-meter track and the same track is returned around it. The researcher will record the distance the patient walks in 6 minutes in meters. The test will be performed in a 60-meter long hospital corridor.

SECONDARY OUTCOMES:
Bristol Breastfeeding Assessment Scale; | 1 HOUR
  "Bristol Breastfeeding Assessment Scale (BEDÖ) was developed by Jenny Ingram in 2014 and adapted to Turkish by Dolgun and her friends in 2017 . The scale was developed to evaluate breastfeeding problems and adequacy encountered frequently in the postpartum period. The mother is observed by a health professional during breastfeeding and the form is filled out by evaluating the mother and the baby in line with the criteria. The application time of the scale is 5-10 minutes. While the Cronbach's Alpha value of the original form of the tool was found to be 0.68, it was found to be 0.77 in the Turkish adaptation study. The measurement tool is a Likert-type scale consisting of 4 items: "positioning", "holding", "sucking" and "swallowing".
  Positioning/Holding: The baby should be well supported, leaned against the mother's body, laid on its side and its neck should not be bent. The nose should be opposite the nipple, the mother sho

IPD SHARING:
Plan to Share IPD: No